CLINICAL TRIAL: NCT06286514
Title: Food at Home Study
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00019996
Record Dates: First submitted 2023-11-29; First posted 2024-02-29 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Obesity; Diet, Healthy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Paper Validation: validate the paper version of the Home Food Inventory
  Interventions: Other: No intervention
- electronic validation: validate the electronic version of the Home Food Inventory
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study

SUMMARY:
The study objective is to develop an accessible home food environment assessment toolkit that includes valid and reliable paper and electronic tools targeting foods known to impact diet-related health that can be user-administered across literacy levels in English and Spanish.

ELIGIBILITY:
Inclusion Criteria:

* Speak Spanish or English at home
* 18 or older
* primary grocery shopper or meal preparer

Exclusion Criteria:

* Any person younger than 18
* lacks the capacity to consent
* does not purchase the majority of the groceries for the home

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 18 who speak either English or Spanish at home and who are responsible for the majority of the cooking or grocery shopping for their family. There will be 150 participants in the paper validation phase (75 who speak English at home and 75 who speak Spanish at home) and 200 participants in the validation of the electronic Home Food Inventory (eHFI) (100 who speak Spanish at home and 100 who speak English at home)
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Usability of HFI core | 1 month
  Primary participant tool completion time
Acceptability of HFI core | 1 month
  Primary participant satisfaction ratings of tool
Concurrent criterion validity of HFI core | 1 month
  Correlations of average HFI-core fruit and vegetable category availability scores between staff (gold standard) and primary participant completed tools
Concurrent criterion validity of HFI core | 1 month
  Correlations of average HFI-core obesogenic scores between staff (gold standard) and primary participant
Convergent construct validity of HFI core | 1 month
  Correlations of participants' average fruit and vegetable category availability scores from HFI core with participants' average corresponding servings of fruit and vegetables reported from average of two days of dietary recall (in native language)
Convergent construct validity of HFI core | 1 month
  Correlations of participants' average obesogenic food availability scores from HFI core with participants' BMI values
Test-retest reliability of HFI core | 1 month
  Correlation coefficient between participants' HFI obesogenic scores from HFI core at visit 1 and visit 2
Usability of eHFI | 1 month
  Primary participant tool completion time
Acceptability of eHFI | 1 month
  Primary participant satisfaction ratings of tool
Concurrent criterion validity of eHFI | 1 month
  Correlations of average eHFI fruit and vegetable category availability scores between staff (gold standard) and primary participant completed tools
Concurrent criterion validity of eHFI | 1 month
  Correlations of average eHFI obesogenic scores between staff (gold standard) and primary participant
Convergent construct validity of eHFI | 1 month
  Correlations of participants' average fruit and vegetable category availability scores from eHFI with participants' average corresponding servings of fruit and vegetables reported from average of two days of dietary recall (in native language)
Convergent construct validity of eHFI | 1 month
  Correlations of participants' average obesogenic food availability scores from eHFI with participants' BMI values

CONTACTS AND LOCATIONS:
Overall Officials: Jayne Fulkerson, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States